CLINICAL TRIAL: NCT01997112
Title: PAracetamol Treatment in Hypertension: Effect on Blood Pressure (PATH-BP) Study
Acronym: PATH-BP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other); National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PATHBP_2013; PG/13/26/3012 8 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Blood Pressure
Keywords: Blood pressure; Hypertension; Paracetamol; Acetaminophen
MeSH Terms: conditions — Hypertension | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paracetamol (Active Comparator): paracetamol 1g (500mg x2) four times daily for 14 day period
  Interventions: Drug: Paracetamol
- Placebo (Placebo Comparator): Matched placebo control: hard gelatin placebo capsules containing Lactose Ph Eur. Taken for 14 days
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Paracetamol
  Other Names: Acetaminophen
  Arms: Paracetamol
Drug: Placebo oral capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine if chronic paracetamol dosing increases blood pressure in patients with known high blood pressure.

DETAILED DESCRIPTION:
A prospective randomised, double-blind, crossover trial, comparing the effects of paracetamol 1g (500mg x2) four times daily with matched placebo on ambulatory and clinic BP, each given for 14 days, with a 14-day washout period.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old, men or post-menopausal women (women with no periods for 12 months or more, or those who have had a surgical menopause)
* Treated hypertensive patients with an average daytime ambulatory blood pressure measurement (ABPM) <150/95mmHg on stable doses of one or more antihypertensive medication (at least one of which should be; an ACE inhibitor, angiotensin receptor blocker or diuretic) for 3 months, or untreated hypertensive patients with an average daytime ABPM ≥135/85 but <150/95.

Exclusion Criteria:

* History of ischaemic heart disease, cardiac failure, cerebrovascular disease, liver impairment (ALT/AST>50IU/L) or stage 3-5 chronic kidney disease.
* History of overdose or suicidal ideation
* Patients weighing <55kgs.
* Patients with chronic pain requiring treatment, with a known allergy to paracetamol, or concomitant use of non-steroidal anti-inflammatories , oral anticoagulants or corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2019-06-04 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Systolic ambulatory blood pressure | 14 days
  Difference in mean daytime systolic ambulatory BP between the paracetamol and placebo treated groups.

SECONDARY OUTCOMES:
Systolic clinic blood pressure | 14 days
  Difference in systolic clinic BP between the paracetamol and placebo treated groups.
Diastolic ambulatory blood pressure | 14 days
  Difference in mean daytime diastolic ambulatory BP between the paracetamol and placebo treated groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Centre, Western General Hospital, Edinburgh, City Of Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] MacIntyre IM, Turtle EJ, Farrah TE, Graham C, Dear JW, Webb DJ; PATH-BP (Paracetamol in Hypertension-Blood Pressure) Investigators*. Regular Acetaminophen Use and Blood Pressure in People With Hypertension: The PATH-BP Trial. Circulation. 2022 Feb 8;145(6):416-423. doi: 10.1161/CIRCULATIONAHA.121.056015. Epub 2022 Feb 7. PMID 35130054